CLINICAL TRIAL: NCT05792241
Title: Evaluation of the Acceptability and Nutritional Impact of Double-fortified Salt Containing Folic Acid and Iodine Among Ethiopian Women of Reproductive Age - Assessment of Women's Nutritional Status and Salt Intakes in the Study Communities
Brief Title: Acceptability and Nutritional Impact of Double-fortified Salt Containing Iodine and Folic Acid - Phase 1
Acronym: DFS-IoFA-1
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Collaborators: Ethiopian Public Health Institute (Other Government); University of California, San Francisco (Other); Nutrition International (Other)
Responsible Party: Sponsor
Other Study IDs: 1834465
Record Dates: First submitted 2023-03-03; First posted 2023-03-31 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Folate Deficiency; Iodine Deficiency; Anemia, Macrocytic; Anemia Deficiency; Salt Intake
Keywords: Ethiopia; Salt fortification
MeSH Terms: conditions — Folic Acid Deficiency; Anemia, Macrocytic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Samples of whole blood, serum, and 24-hour urine excretion will be collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women of reproductive age: Randomly selected women of reproductive age in study communities.

SUMMARY:
The overarching objective of this two-phase project is to assess the effects of fortifying iodized salt with folic acid on improving women's folate status and thereby reduce the risk of neural tube defects (NTDs), which are highly prevalent in Ethiopia. The project will be conducted in two phases. The purpose of Phase 1, described herein, is to complete formative research in preparation for a community-based, randomized trial, which will be carried out in Phase 2. The objectives of Phase 1 are to: 1) assess the hematological condition and nutritional status with respect to folate, iodine, and other micronutrients among non-pregnant women of reproductive age (WRA) in the study communities, and 2) measure discretionary salt and dietary folate intakes of the women and their households.

DETAILED DESCRIPTION:
Potentially eligible women of reproductive age (WRA) will be identified from existing community census records and will be listed sequentially. A random number generator will be used to select individual women from this list for possible participation in the Phase 1 studies. In cases where two or more WRA are selected from the same household (HH), one will be randomly selected for possible participation in the study and the other(s) will be replaced by a WRA from another HH, using the same random selection procedure. A member of the study team will then visit the homes of women who are selected for possible participation in Phase 1 to describe the study to them, assess their eligibility, and request their consent to participate. In particular, the data collector will present an initial disclosure statement concerning the screening interview and will then obtain descriptive information from verbally consenting women on their age, general health status, address, cell phone number (if available), and potential willingness to participate in the subsequent research studies. The data collector will review the women's health history and determine their eligibility for the Phase 1 study.

For women who found to be eligible to participate in the Phase 1 study, the field worker will describe the purpose of the study, the study procedures and related risks and benefits, the confidentiality of results, and the fact that participation is voluntary. After providing an opportunity for women to consult with family members and ask any questions to the research team, the field worker (in the presence of a neutral witness) will request written consent from the women to participate in the study. Additional questions will be asked of consenting women regarding their marital status, ethnicity, religion, educational level, and employment; and their housing characteristics (housing construction, water source, sanitary facilities, access to electricity and cell phone service); and selected HH assets.

All eligible, consenting women will be requested to report to the Chefe Donsa Health Center or one of the local health posts within the next one or two days following the initial screening interview for fasting blood collection, anthropometric assessment, additional interviews, and scheduling of subsequent home visits by the study team for full-day dietary observations to measure discretionary salt intake and folate intake and to initiate 24-hour urine collections to measure sodium and iodine excretion. The fasting blood specimens will be collected for a complete blood count and measurement of red blood cell (RBC) folate and serum folate, unmetabolized folic acid, vitamin B12, holo-transcobalamin, methyl malonic acid, other B vitamins, genetic polymorphisms that affect folate metabolism, thyroglobulin, glucose, insulin, retinol binding protein (RBP), ferritin, soluble transferrin receptor, C-reactive protein, and alpha-1 acid glycoprotein and to complete a malaria rapid diagnostic test (RDT). Serum retinol will be measured in a subset of 40 women to establish the relationship between serum retinol and RBP in the study population. Blood specimens may also be collected from a subset of 20 women for possible metabolomics assays and natural killer cell (immune function) assays. Women with a positive RDT and those subsequently found to have anemia (Hb<13.2 g/dL, to adjust for altitude) will be referred to the local health facility for treatment. Additional interviews will be completed to assess the women's birth history, contraceptive use, and household food insecurity.

All women will participate in dietary assessments and 24-hour urine collections on one day within four weeks of enrollment, and a randomly selected sub-set of 40 women will complete these studies on a second day one-to-two weeks later. The purpose of the second set of studies is to allow for calculation of intra-individual variation in intakes and urinary sodium and iodine excretion, which is necessary to estimate the distribution of usual discretionary salt and folate intake and urinary sodium and iodine excretion of the study population. The dietary studies will involve a dietitian who will remain in the participant's home throughout the day to weigh all foods included in mixed dishes and to weigh the amounts served and consumed. Portions of each food will be collected to analyze these in the laboratory for sodium and selected nutrient contents. The investigators The investigators will also carry out HH salt disappearance studies over a period of one week using iodized refined salt provided by the project to determine the rate of salt utilization in relation to HH size. This information will be used to estimate the quantities of salt that we will need to deliver during Phase 2.

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant women 18-49 years of age
* Agree to use salt provided by the study team for the household salt disappearance study
* Provide written, informed consent.

Exclusion Criteria

* Currently pregnant
* Presence of acute or chronic disease (such as diarrhea, febrile illness, or underlying metabolic disorder) that might affect the participant's dietary intake or folate status
* Currently using medicines (like anticonvulsants and cancer treatments) that affect folate metabolism
* Medically prescribed restriction of salt intake

Ages: 18 Years to 49 Years | Sex: Female
Age Groups: Adult
Study Population: The study will be conducted in the central highlands of Oromia region in Ethiopia, approximately 2 hours from the capital Addis Ababa.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-06-26 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Folate status | one week
  Red blood cell (RBC) folate concentration using a microbiological assay
Iodine status | four weeks
  24-hour urinary iodine excretion using the Sandell-Kolthoff color reaction
Discretionary salt intake | four weeks
  In-home weighed record of dietary intake
Household salt utilization | six weeks
  One-week difference in weight of salt provided by study team

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth H Brown, MD, Principal Investigator — University of California, Davis
Locations (1):
- Ethiopian Public Health Institute, Addis Ababa, Ethiopia

IPD SHARING:
Plan to Share IPD: Yes
Two years after completion of the data collection, the individual participant data (IPD) data sets will become publicly available to other investigators who have specific research questions that can be addressed by the data and that are not already under analysis by the core research team. Researchers who desire to have access to the clinical specimens will be requested to apply for the specimens and to describe the research question(s) they plan to address.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The study protocol will be submitted for publication prior to initiation of Phase 2. The statistical analysis plans for Phases 1 and 2 will be publicly available prior to the start of the respective analyses. The informed consent documents will be available (in English and Afaan Oromo) after approval by the respective institutional Review Boards (IRBs) at the University of California Davis (UC Davis) and the Ethiopian Public Health Institute (EPHI). The clinical study report will become available once accepted for publication.
Access Criteria: As indicated above.

REFERENCES:
- [Result] Agbemafle I, Woldeyohannes M, Tessema M, Fereja M, Arnold CD, Banjaw BT, Hussen A, Kebebe T, Goh YE, Arabi M, Martinez H, McDonald CM, Brown KH. Assessment of Women's Discretionary Salt Intake and Household Salt Utilization in Preparation for a Salt Fortification Trial in Oromia Region, Ethiopia. Matern Child Nutr. 2025 Apr;21(2):e13768. doi: 10.1111/mcn.13768. Epub 2024 Dec 13. PMID 39673143